CLINICAL TRIAL: NCT03241433
Title: High-Intensity Interval Training and Moderate-Intensity Continuous Training in Reducing Atrial Fibrillation Burden
Brief Title: High-Intensity Aerobic Lifelong Training--AF
Acronym: HALT-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1703M11461
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Atrial Fibrillation
Keywords: Exercise
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity interval training (Active Comparator): Exercise training will be conducted 3 times per week using cycle ergometers at commercial fitness facilities for 12 weeks 2 minute warmup/3 minute cooldown- at 50W Intensity- 3 X 20-second sprint interval cycling -as fast as possible at 90-95% peak power low intensity- 2 X 2 minute cycling at slow pace 50W
  Interventions: Other: High intensity interval training
- Moderate intensity continuous training (Active Comparator): Exercise training will be conducted 3 times per week using cycle ergometers at commercial fitness facilities for 12 weeks 2 minute warmup/3 minute cooldown- at 50W Intensity- 45 minutes of continuous cycling at 45-60% peak power
  Interventions: Other: Moderate intensity continuous training
- No exercise (Active Comparator): No excercise training will be done
  Interventions: Other: No Exercise

INTERVENTIONS:
Other: High intensity interval training — exercise by use of stationary cycles
  Arms: High intensity interval training
Other: Moderate intensity continuous training — exercise by use of stationary cycles
  Arms: Moderate intensity continuous training
Other: No Exercise — no exercise training will be given and no exercise will be added to subjects routine
  Arms: No exercise

SUMMARY:
This study is a single-center RCT. Potential subjects with symptomatic non-permanent AF will be enrolled to determine the effect of sprint interval training (SIT) in comparison to moderate-intensity continuous training (MICT) and non-exercise control in reducing AF burden. The Investigators will enroll 60 patients during the first 12 months of the study. Baseline data collection will be conducted during the first month after enrollment. After baseline data collection, subjects will be randomized (1:1:1) to SIT vs. MICT vs. non-exercise controls. The exercise training will last for 3 months followed by final data collection which will be completed in 1 month.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm abnormality in the general population. Current recommended methods to maintain sinus rhythm or reduce AF burden (% time a person is in AF) in patients with non-permanent AF are costly and ineffective. Hence, there is an urgent need to discover novel inexpensive strategies to reduce AF burden. It is well-established that regular aerobic exercise reduces cardiovascular morbidity and mortality; however, adherence to regular exercise is poor rendering it an ineffective public health strategy. Evidence is emerging to suggest that traditional moderate-intensity continuous training (MICT) and high-intensity interval training (HIIT) may be associated with lower AF burden. Compared with traditional MICT, HIIT is possibly more time-efficient; hence, it may promote adherence. Since lack of time is the most common reason for poor adherence to regular exercise, the time-efficiency of HIIT holds promise to be a "game-changer". However, many knowledge gaps remain. First, HIIT has never been compared directly with MICT in relation to AF burden; thus, whether HIIT is comparable or superior to MICT is unknown. Second, the time commitment required for a "conventional" HIIT program (120 mins/week) is not substantially less than the recommended MICT (150 mins/week); hence, it is doubtful that it can be a real "game-changer" in terms of promoting adherence. Third, HIIT performed using a cycle ergometer is a safer alternative to the treadmill in older adults, but has not been evaluated in patients with AF. Finally, mechanisms underlying the salutary benefits of exercise in relation to AF burden remain unknown. To address these knowledge gaps, the investigators will evaluate an innovative HIIT program-sprint interval training (SIT)-using a cycle ergometer that only requires 10 minutes per session and 30 minutes per week, in contrast to the "conventional" HIIT program that requires 40 minutes per session and 120 minutes per week. In this pilot randomized controlled trial (RCT), the investigators will randomize 60 subjects with non-permanent AF (1:1:1) to SIT vs. MICT vs. no exercise control. At enrollment, these subjects will undergo heart rhythm monitoring by a non-invasive ambulatory heart rhythm monitor, V02 max testing, assessment of cardiac size and function by cardiac MRI, and assessment of AF symptom severity; these measures will be repeated at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* : Patients with symptomatic non-permanent AF and aged 18-65 years who are sedentary (activity ≤0.5 hours/week of regular exercise) and seen by Dr. Chen or his cardiology colleagues at Clinics and Surgery Center (CSC), other Fairview cardiology clinics, and University of Minnesota Medical Center (UMMC). Patients will be screened and enrolled by a research coordinator.

Exclusion Criteria:

* Individuals lacking the capacity to consent for themselves will not be included, previous open heart surgery, previous catheter ablation for AF, LVEF <45%, significant cardiac valve disease, coronary heart disease without complete revascularization, implanted cardiac electronic device, or GFR <30 mL/min/1.73 m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Change in AF burden | 3 months
  After 12 weeks of exercise training , HIIT and MICT will be comparable but better than non-exercise control in AFburden(% of time a person is in AF) by using an ambulatory patch monitor

SECONDARY OUTCOMES:
Change in left atrial and left ventricular size and function | 3 months
  After 12 weeks of exercise training HIIT and MICT will be comparable but better than non-exercise control as Cardiac MRI will be completed to assess LV and LA volumes and function and LV fibrosis
change in clinical outcomes | 3 months
  The favorable effect of HIIT and MICT over non exercise control on clinical outcomes will be attenuated after after for secondary outcomes, suggesting that the latter mediate the clinical benefits of regular aerobic exercise

CONTACTS AND LOCATIONS:
Overall Officials: Lin Yee Chen, MD,MBBS,MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No